CLINICAL TRIAL: NCT04948164
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of the Efficacy and Safety of Sumatriptan Naproxen Sodium Succinate Tablets for the Treatment of Acute Migraine Attacks.
Brief Title: Study of Sumatriptan Naproxen Sodium Succinate Tablets for the Treatment of Acute Migraine Attacks
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Second Hospital of Jilin University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); The Second Hospital of Nanjing Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Beijing Friendship Hospital (Other); West China Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2018061
Record Dates: First submitted 2021-06-27; First posted 2021-07-01 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Migraine in Adults
MeSH Terms: interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Drug: sumatriptan 85mg and naproxen sodium 500mg
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sumatriptan 85mg and naproxen sodium 500mg — Subjects took 1 tablet of the study drug (each containing sumatriptan 85mg and naproxen sodium 500mg) within 1h of an acute migraine attack of mild severity, and if the headache progressed to moderate severity within 2 hours, they could take the remedial drug phenol chai (each containing acetaminophen 500mg and caffeine 65mg).
  Arms: Test group
Drug: Placebo — subjects were given one tablet of placebo within 1 h of an acute migraine attack with mild severity, and if the headache progressed to moderate severity within 2 hours, they were given the remedial drug phenol chai (each tablet contains acetaminophen 500 mg and caffeine 65 mg)."
  Arms: Control group

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of sumatriptan naproxen sodium succinate tablets in the treatment of acute migraine attacks.

DETAILED DESCRIPTION:
Migraine is a common chronic nerve vascular disease, the disease characteristic to break out repeatedly, one side or both sides of the pulsatile partial side head, severe headache and can combine autonomic nervous system dysfunction such as nausea, vomiting, photophobia, and fear the symptom such as, about one-third of patients with migraine aura symptoms can appear before the onset of the nervous system. Sulaptan is a 5-HT1 receptor agonist with a high affinity for binding to 5-HT1b and 5-HT1D receptors. Naproxen is an NSAID that inhibs the synthesis of inflammatory mediators. Thus, sulaptan and naproxen alleviate migraine through different pharmacological mechanisms of action. For this test center, randomized, double-blind, placebo-controlled, parallel-group Ⅲ phase of clinical trial, aimed to verify shu Ma Putan naproxen sodium treatment of acute migraine headache, headache complete remission rate after 2 hours, evaluation of succinic acid shu Ma Putan naproxen sodium tablets for efficacy and safety of the treatment of acute migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old and <65 years old at the time of signing the informed consent form, regardless of gender;

  2. Diagnose patients who meet the criteria for the diagnosis of migraine without aura in the third trial version of the International Classification of Headache Diseases (ICHD-Ⅲ(β)) launched by the International Headache Association, and the degree is moderate or severe;

  3. The age of the patient's first migraine attack should be less than 50 years old, and must meet 5 or more migraine attacks without aura or a history of migraine without aura ≥ 1 year;

  4. The number of moderate or severe migraine attacks ≤6 and ≥1 per month within the first 3 months of enrollment, and at least a 48-hour headache interval;

  5. Ability to distinguish migraine patients from other types of headaches during headache attacks;

  6. Female patients who have not had unprotected sex in the 15 days before screening, and patients (regardless of men and women) who have no childbirth plans during the trial period and within 6 months after the end of the trial;

  7. Patients who have the ability to cooperate in observing curative effects and adverse events, and record headache diaries;

  8. Before starting any detailed procedures of this study, the patient has the ability to understand and sign a written informed consent form approved by the ethics committee

Exclusion Criteria:

* 1. Patients with migraine with aura, including but not limited to patients with brainstem migraine with aura and patients with hemiplegic migraine;

  2. Patients with average headache time ≥15 days per month in the 3 months before the test;

  3. Patients who have taken painkillers for a long time or overuse of painkillers (take painkillers for more than 10 days a month for 3 consecutive months);

  4. Abnormal renal function: creatinine value> upper limit of normal value;

  5. Patients with a history of severe liver disease or patients with significantly abnormal liver function: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≥ 1.5 times the upper limit of normal or total bilirubin (TBIL) )≥1.5 times the upper limit of the normal value;

  6. History of major mental and neurological diseases such as depression and epilepsy;

  7. Patients who have taken central sedatives for a long time, such as barbiturates and benzodiazepines, including diazepam, lorazepam, etc.;

  8. Patients with severe cardiovascular diseases, such as coronary artery bypass surgery, or patients with a history of one of the following diseases, including but not limited to ischemic heart disease, such as angina (including Platts variant angina), Patients with a history of myocardial infarction, arrhythmia (such as pre-excitation syndrome) or disease-related symptoms, signs, or a significant ECG abnormal change;

  9. Patients with severe cerebrovascular diseases, including but not limited to cerebral ischemia, cerebral hemorrhage diseases;

  10. With severe peripheral vascular disease, such as Raynaud's syndrome;

  11. Patients whose blood pressure cannot be effectively controlled after drug treatment, systolic blood pressure (SBP)>140mmHg or diastolic blood pressure (DBP)>90mmHg;

  12. Take ergotamine or ergot derivatives (such as dihydroergotamine or ergonovine) or other 5-HT1 receptor agonists within 7 days before randomization;

  13. Patients who have taken MAOI within 14 days before screening;

  14. Patients who cannot stop using anticoagulant drugs (such as warfarin) or antiplatelet drugs (such as aspirin) during the trial;

  15. Patients who have previously undergone gastric resection or bypass surgery, or patients with a history of gastrointestinal bleeding, ulcers, or perforation;

  16. Patients suffering from sinusitis;

  17. Regularly take drugs for preventing headache attacks for more than 2 weeks before randomization, including but not limited to flunarizine, topiramate and Chinese patent medicines with similar effects;

  18. Known to triptan drugs, NSAIDs or their pharmaceutical excipients Patients with allergies, or have had aspirin asthma or aspirin triad (aspirin allergy, asthma, and nasal polyps);

  19. For patients with alcohol abuse and drug abuse, the standard for alcohol abuse is: drinking an average of more than 28 units per week (a unit of alcohol is equivalent to 250 mL of beer, 125 mL of wine or 20 mL of spirits or enthusiastic alcoholism); There are two types of drugs: one is narcotic drugs, such as heroin, marijuana and cannabis resin, opiates and morphine preparations, codeine, etc.; the other is psychotropic drugs, such as various hallucinogens and tetrahydrocannabinol, central stimulants Drugs, barbiturates, benzodiazepines, etc.;

  20. Patients who are pregnant, breastfeeding, or have a childbearing plan during the study period, including female patients of childbearing age who have a positive pregnancy test;

  21. Patients who have participated in any other clinical trials within 3 months before participating in this trial, and who plan to participate in other clinical trials of other drugs;

  22. The patient may not be able to complete the trial due to reasons, or the investigator believes that the patient is not suitable to participate in this trial. "

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Relief rate | 2hr after taking the drug
  Complete headache relief rate within 2 hours after taking the drug for the first time (proportion of subjects without headache)

CONTACTS AND LOCATIONS:
Overall Officials: Yingshuang Zhang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No